CLINICAL TRIAL: NCT06215638
Title: An Exploratory Clinical Study on Bortezomib for the Treatment of Refractory Rheumatoid Arthritis
Acronym: bortezomib4ra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-23PJ350
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; Bortezomib; difficult-to-treat rheumatoid arthritis; refractory rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 2 mg per week subcutaneously, for twelve weeks in total

SUMMARY:
The goal of this prospective single-arm open-label trial is to learn about efficacy and safety of Bortezomib in treating patients with difficult-to-treat rheumatoid arthritis. The main questions it aims to answer are:

* Is Bortezomib an effective treatment option for patients with difficult-to-treat rheumatoid arthritis?
* Is Bortezomib safe enough in treating patients with difficult-to-treat rheumatoid arthritis?

Participants will:

* Receive Bortezomib 2 mg per week subcutaneously for twelve weeks in total.
* Follow-up at weeks 4, 12, and 24, while biosamples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <70 years;
* Absolute neutrophil count ≥1.0×10^9/L, platelet count ≥100×10^9/L, aspartate transaminase and total bilirubin within 3 times and 1.5 times the normal upper limit, respectively, and serum creatinine clearance >60 ml/min;
* Voluntarily sign an informed consent form.

Exclusion Criteria:

* Individuals with concomitant autoimmune diseases;
* Presence of severe, poorly controlled cardiovascular, cerebrovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neuropsychiatric diseases, or laboratory abnormalities that the investigator deems an unacceptable risk for the participant's involvement in the study;
* History of malignant tumors (or clinical cure time less than 5 years);
* Subjects who are pregnant or lactating, or planning to become pregnant or start breastfeeding during the study period;
* Vaccination with live virus vaccines within the 4 weeks prior to study entry;
* Allergy to Borussertib or mannitol;
* Participation in any other investigational drug trial in the 12 weeks before the start of this study medication;
* Presence of active hepatitis or a history of severe liver disease at screening: defined as a positive test for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus antibodies (HCVAb) (Note: If the result of hepatitis B core antibody (HBcAb) is positive and HBsAg is negative, hepatitis B virus (HBV) DNA testing will be performed. If HBV-DNA is negative, the patient is eligible.);
* Active herpes zoster infection, or occurrence of a severe infection in the 12 weeks before the start of the study medication (defined as requiring intravenous antibiotics or hospitalization);
* Other situations that investigators deem unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
ACR20 | From enrollment to week 12
  The ACR response criteria for 20 percent improvement in disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical Cllege Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No